CLINICAL TRIAL: NCT04144062
Title: CAD/CAM Crowns Versus Prefabricated Zirconia and Stainless Steel Crowns for Restoration of Primary Molars: A Prospective Study.
Brief Title: Primary Molars Restoration Using Different Pediatric Crowns.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nehal Salman (Other)
Responsible Party: Sponsor-Investigator, Nehal Salman, Lecturer, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 318
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2021-02

CONDITIONS: Restoration of Primary Molars With CAD/CAM Crowns
Keywords: Crowns; Zirconium; Computer-Aided Design

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Zirconia crowns (Active Comparator)
  Interventions: Other: CAD/CAM crowns
- CAD/CAM crowns (Active Comparator)
  Interventions: Other: CAD/CAM crowns
- Stainless-steel crowns (Active Comparator)
  Interventions: Other: CAD/CAM crowns

INTERVENTIONS:
Other: CAD/CAM crowns — CAD/CAM crowns

SUMMARY:
study aims to compare hybrid ceramic CAD/CAM and prefabricated zirconia ans stainless steel crowns restoring primary molars through In-vivo evaluation of the clinical outcomes in terms of; crown retention, stain resistance and periodontal and gingival health as well as parental/child satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of the patients from 5 to 8 years old.
2. Have no history of spontaneous pain or swelling.
3. Patients willing to return for follow-up examinations and evaluation.
4. Medically free patients or with controlled systemic disease ASA I or II.
5. No active periodontal diseases.
6. Patients with posterior pulpotomized tooth/teeth indicated for crown restoration (e.g. 2-3mm of teeth above cement-enamel junction).

Exclusion Criteria:

1. Children with intellectual, severe emotional or behavioral problems.
2. Presence of parafunctional habits such as clenching or bruxism.
3. Abnormal tooth mobility, gingival swelling, fistulous tract, or non-vital pulps.
4. Non-restorable teeth.
5. Radiographic positive signs of thickened or interrupted periodontal membrane space, internal root resorption, periapical or furcal radiolucency

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
clinical success | 1 year
  United States Public Health Service (USPHS) index

CONTACTS AND LOCATIONS:
Locations (1):
- Nehal Salman, Alexandria, Egypt, Egypt